CLINICAL TRIAL: NCT00873184
Title: Feasibility Study of Massage Therapy Within a Brain Tumor Setting
Brief Title: Study of Massage Therapy Within a Brain Tumor Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Massage Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010000
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2012-03

CONDITIONS: Brain Tumors
Keywords: massage therapy in patients with brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): A prospective, single-arm intervention study, potential participants will be identified and screened for eligibility via medical record review of patient scheduled for their post surgical primary adjuvant treatment consultation at DUMC.
  Interventions: Behavioral: Massage Therapy

INTERVENTIONS:
Behavioral: Massage Therapy — The setting for massage intervention will take place at The Duke Center for Living (DCL). . The massage therapists at the DCL work closely with physicians to design appropriate interventions for patients who are receiving treatment at DUMC, including cancer patients. All DCL therapists have completed more than 600 hours of training, are nationally certified and hold a North Carolina license to practice massage. These types include Swedish, deep muscle, myofascial release, trigger point, acupressure, Bowen Technique, sports massage and chair massage.

SUMMARY:
The purpose of this study is

* to assess the feasibility and acceptability of massage therapyto examine the effects of massage therapy
* to explore whether psychological outcomes are associated with changes in patient reported QoL.

DETAILED DESCRIPTION:
As a part of this study, we will provide massage therapy to brain tumor patients. Our contribution here is expected to determine whether massage therapy is safe and helps to improve patient QoL. This contribution is significant because it is expected to provide pilot data on effect sizes so that we may design an adequately powered study to develop massage therapy programs and interventions for patients with brain tumors. In addition to benefiting brain tumor patients, the information from this study may be applied to improving the QoL of other cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmed, newly diagnosed, post surgical WHO grade III/IV malignant glioma (i.e., glioblastoma, anaplastic astrocytoma) being followed at the Preston Robert Tisch Brain Tumor Center (PRT-BTC) at Duke University Medical Center (DUMC) will be considered potential participants for this study.
* Additional eligibility criteria will be:

  1. > 18 years old
  2. Karnofsky Performance Score of > 70 at onset of study
  3. estimated life expectancy of > 3 months
  4. approval from attending oncologist
  5. the ability to speak, read and write English
  6. live within a 60 mile radius of the DCL
  7. be identified as "stressed" by Perceived Stress Scale (PSS) score, > 12.1 and 13.7 for men and women respectively, and 8) signed informed consent prior to initiation of study-related procedures.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility and acceptability of massage therapy provided to primary brain tumor patients. This assessment will integrate data about patient eligibility rates, patient participation rates, patient adherence rates, and adverse events. | 6 months

SECONDARY OUTCOMES:
To examine the effects of massage therapy on psychological outcomes related to stress, distress, anxiety, and depression in this population and to explore whether psychological outcomes are associated with changes in patient reported QoL. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Keir, Dr.Ph,MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States